CLINICAL TRIAL: NCT01922934
Title: A Toolbox Approach to Obesity Treatment in Primary Care
Acronym: Toolbox
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Daniel Bessesen, Principal Investigator, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GM3469
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Phentermine; Qsymia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 350 randomly-selected patients at 4 clinics get a "toolbox" of weight loss options, including self-monitoring tools; education materials; recreation center passes; commercial weight loss program (Weight Watchers); intensive group counseling (Colorado Weigh); meal replacements; and obesity pharmacotherapy. The initial assessment, a computer program, takes diet and exercise history and helps patients choose personal treatment goals. Interested patients get a starter kit with self-monitoring tools and meal replacements. Subjects must show self-monitoring of diet and exercise to get more intensive therapies. Patients pay a $5-$10 co-pay for the therapies. They select a primary intensive therapy, but are able to add/change depending on results, adherence and budget availability.
  Interventions: Behavioral: Commercial weight loss program; Behavioral: Colorado Weigh; Dietary Supplement: Meal replacements; Drug: Obesity pharmacotherapy; Behavioral: Recreation center passes
- Control (No Intervention): Registry patients not selected to be offered the toolbox will receive usual care for weight management. Usual care for obesity at DH includes brief weight loss advice provided by PCPs or prescribing of weight loss medication, for which patients pay out of pocket.

INTERVENTIONS:
Behavioral: Commercial weight loss program — vouchers for Weight Watchers
  Arms: Intervention
Behavioral: Colorado Weigh — Group behavioral weight loss program
  Arms: Intervention
Dietary Supplement: Meal replacements — Health Management Resources meal replacement products (shakes and entrees)
  Arms: Intervention
Drug: Obesity pharmacotherapy — Phentermine or phentermine-topiramate (Qsymia)
  Other Names: Phentermine or phentermine-topiramate (Qsymia)
  Arms: Intervention
Behavioral: Recreation center passes — 1 year pass to a Denver recreation center
  Arms: Intervention

SUMMARY:
Obesity is common, causing many medical problems in adults (e.g., diabetes, hypertension, high cholesterol, sleep apnea, heart attack, strokes). A range of treatments have shown to be effective for treating obesity. Treatments include lifestyle modification, meal replacements, and weight loss medication. Most primary care settings do not provide much obesity treatment, though, as primary care providers (PCPs) are not well trained and because reimbursement for treatments is not consistent.

Hypothesis: If PCPs have training in weight management and if most costs of treatment are reimbursed, we surmise that a "toolbox" of treatments can produce a clinically important weight loss amount in a large group of patients.

Design: We propose to establish a registry of obese patients with at least one common medical condition related to their weight. From the registry, we will randomly select 350 people to be offered treatments to assist with weight loss. The remainder of the registry's patients can still receive obesity treatment but will not be reimbursed. We will conduct the study at Denver Health, a large public health care system that treats a low income, ethnically diverse population. All 350 patients will be offered some self-monitoring tools for weight management and the chance to do a computer assessment to select the right treatment for weight loss. Patients who complete this and record their food intake and physical activity for 1 week will be offered a "Level 2" treatment for weight loss. Level 2 treatments include: a voucher for a commercial weight loss program; intensive group weight loss counseling; meal replacements; gym membership; or weight loss medication. Patients will choose which treatment they want, with the approval of their PCP. Researchers at Denver Health will help with the computer assessment and dispensing the treatments. We are interested in what percentage of patients lose at least 5% of their starting weight. We will also explore changes in glucose, blood pressure, and cholesterol, and we will look at how much this intervention costs and whether patients need less medication for their weight-related conditions at the end of the study.

Impact: If the study is successful, we plan to take the results to the leaders at Denver Health to see if they will make obesity treatment more broadly available for all patients there.

DETAILED DESCRIPTION:
Background: Obesity is prevalent and is a root cause of many common medical conditions affecting U.S. adults. A range of treatment options have demonstrated efficacy in producing weight loss and reducing health risks in randomized controlled trials. However, very little obesity treatment is currently delivered in most primary care settings. Inadequate reimbursement for treatment modalities and a lack of systematic training of primary care providers (PCPs) are two of the major barriers to more widespread treatment.

Hypothesis: If PCPs are given training and support for weight management, and if treatment options with proven efficacy are offered to obese adults with weight related co-morbidities with the majority of the treatment cost reimbursed, then clinically meaningful weight loss will be produced in a significant number of these individuals at a reasonable cost.

Design: This application proposes a 12 month intervention trial among obese adults cared for at 4 primary care clinics affiliated with Denver Health (DH), an integrated health care system serving an ethnically diverse medically underserved population. From among a large population of patients (~8,000) with obesity and at least one co-morbid condition, 350 individuals will be randomly selected to be offered a "toolbox" of treatment options. The remainder will be assigned to a control condition. The "toolbox" will include: 1) meal replacements; 2) group weight loss counseling; 3) membership at recreation centers; 4) pharmacotherapy with phentermine; and 5) other options. Patients in the intervention arm will undergo an initial evaluation using an "expert systems" computer program. They will then be required to self-monitor diet and physical activity before gaining access to the higher cost weight management services in the toolbox. Primary care providers will help patients choose treatment approaches, encourage adherence, and monitor success. Patient Navigators will assist patients in accessing prescribed treatments. The primary outcome will be the fraction of patients in each group who achieve a 5% weight loss after 12 months of intervention. Secondary outcomes will include uptake and utilization of treatment options, changes in cardiovascular disease risk factors, and other health care utilization, in particular outpatient medications for diabetes, hypertension, and lipids. While the treatment modalities to be used in this trial are not new, an intervention delivering a toolbox of weight management services in a safety net clinical setting and examining the effect on health care utilization is innovative. The submitted letters of support attest to the need for more data so that health care providers and payers can make evidence-based decisions regarding the provision of obesity treatment to large patient populations.

Impact: A positive result would encourage the broader adoption of a toolbox approach to weight management in primary care settings. A negative result would strongly suggest that even with a "best case scenario" of training and support for obesity treatment, the primary care clinic is not an effective route of delivery for weight management. Either result would be important in shaping future policy decisions about obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 30 kg/m2 and < 45 kg/m2
2. Any one of the following (weight-related) diagnoses: type 2 diabetes or pre-diabetes, including those treated with glucose lowering medications; hypertension, including patients treated with anti-hypertensive medications; hyperlipidemia, including those treated with lipid lowering agents; atherosclerotic cardiovascular disease, including coronary heart disease, cerebrovascular disease, or peripheral vascular disease; obstructive sleep apnea
3. Visited their primary care provider (PCP) at least twice during the past 12 months, including once in the last 6 months

Exclusion Criteria:

Heart attack or stroke within the past 6 months; cancer treated within the past 5 years, except for non-melanoma skin cancer or localized prostate cancer; other medical contraindications to weight loss (e.g., end-stage renal disease, cirrhosis); active substance abuse; current treatment for bipolar disorder or schizophrenia; discretion of PCP (see below)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4730 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Bessesen, MD, Principal Investigator — Chief of Endocrinology at Denver Health
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saxon DR, Chaussee EL, Juarez-Colunga E, Tsai AG, Iwamoto SJ, Speer RB, Heyn H, Kealey EH, Bessesen DH. A Toolbox Approach to Obesity Treatment in Urban Safety-Net Primary Care Clinics: a Pragmatic Clinical Trial. J Gen Intern Med. 2019 Nov;34(11):2405-2413. doi: 10.1007/s11606-019-05222-0. Epub 2019 Aug 26. PMID 31485965
- [Derived] Iwamoto S, Saxon D, Tsai A, Leister E, Speer R, Heyn H, Kealey E, Juarez-Colunga E, Gudzune K, Bleich S, Clark J, Bessesen D. Effects of Education and Experience on Primary Care Providers' Perspectives of Obesity Treatments during a Pragmatic Trial. Obesity (Silver Spring). 2018 Oct;26(10):1532-1538. doi: 10.1002/oby.22223. Epub 2018 Sep 26. PMID 30257072

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: 428 randomly-selected patients from four Denver Health clinics are identified for the intervention arm which offers a "toolbox" of weight loss options. The "toolbox" includes: self-monitoring tools; education materials; recreation center passes; commercial weight loss program vouchers (Weight Watchers); intensive group counseling (Colorado Weigh); meal replacements (shakes & entrees); and obesity pharmacotherapy (Qsymia & phentermine). At the initial assessment (visit 0), a computer program helps patients choose a personal treatment mode and they receive a starter kit with self-monitoring tools and meal replacements. Subjects must show self-monitoring of diet and exercise to receive more intensive therapies at their next visit (visit 1). At subsequent monthly visits, patients select a primary intensive therapy, but are able to add/change tools throughout the one year study period. Patients pay a $5-$10 co-pay for the therapies.
- Control: 4302 Registry patients not selected to be offered the "toolbox" options will receive usual care for weight management. Usual care for obesity at DH includes brief weight loss advice provided by PCPs or prescribing of weight loss medication, for which patients pay out of pocket.
Period: Eligible Patients
Arm/Group | Intervention | Control
Started | 428 | 4302
Completed | 375 (375 patients determined eligible after original random selection from DHHA data warehouse.) | 4214 (81 patients did not meet inclusion criteria as they were 80 years or older. 7 patients had died.)
Not Completed | 53 | 88
Not completed — Death | 0 | 7
Not completed — Physician Decision | 17 | 0
Not completed — Did not meet inclusion criteria | 36 | 81
Period: Visit 0 - Patient Contacted & Consented
Arm/Group | Intervention | Control
Started | 375 | 4214 (Control group patients were not contacted or offered intervention)
Completed | 140 (reflects number of patients that were contacted and agreed to attend Visit 0) | 4214
Not Completed | 235 | 0
Not completed — Patient declined to participate | 169 | 0
Not completed — No response or could not reach | 66 | 0
Period: Visit 1- Weight Measured
Arm/Group | Intervention | Control
Started | 140 (21 patients did not return for Visit 1 to receive tool or have weight measured.) | 4214
Completed | 119 (Patients first received tool and were weighed at Visit 1) | 2930 (1284 patients did not have any weights recorded in EMR during study timeframe)
Not Completed | 21 | 1284
Not completed — Did not have weight recorded (visit 1) | 21 | 1284
Period: Visit 12 / Final Visits
Arm/Group | Intervention | Control
Started | 119 | 2930
Completed | 113 (6 patients did not return for final visit and weight measure) | 2640 (290 patients did not have a second weight recorded at one year (+/- 6months) of first weight)
Not Completed | 6 | 290

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Subjects who were offered the toolbox of weight loss interventions and paid at least one co-pay to start using a tool.
- Registry-Based Control Group: Eligible subjects from an obesity registry (i.e. BMI >/= 30 and at least one weight-related comorbidity) who had at least one measured weight during usual care during the 12-month study period.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Registry-Based Control Group | Total
Number analyzed (Participants) | 119 | 2930 | 3049
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 2475 | 2578
  >=65 years | 16 | 455 | 471
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [42 to 60] | 52 [42 to 61] | 52 [42 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 2064 | 2147
  Male | 36 | 866 | 902
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 1859 | 1924
  Not Hispanic or Latino | 54 | 1071 | 1125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 8 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 545 | 565
  White | 98 | 2335 | 2433
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 42 | 42
Baseline BMI [Count of Participants; unit: Participants]
  30-34.9 | 62 | 1612 | 1674
  35-39.9 | 32 | 901 | 933
  40-44.9 | 25 | 417 | 442
Baseline BMI (continuous) [Median (Inter-Quartile Range); unit: kg/m^2] | 34.6 [32.4 to 39.4] | 34.3 [31.9 to 37.7] | 34.4 [31.9 to 37.8]
Primary Language [Count of Participants; unit: Participants]
  English | 84 | 2033 | 2117
  Spanish | 35 | 897 | 932
Diabetes, hypertension, or hyperlipidemia [Count of Participants; unit: Participants]
  Had at least one | 99 | 2376 | 2475
  Have none | 20 | 554 | 574
Diabetes [Count of Participants; unit: Participants]
  Yes | 58 | 1350 | 1408
  No | 61 | 1580 | 1641
Hypertension [Count of Participants; unit: Participants]
  Yes | 78 | 2063 | 2141
  No | 41 | 867 | 908
Hyperlipidemia [Count of Participants; unit: Participants]
  Yes | 63 | 1596 | 1659
  No | 56 | 1334 | 1390
Coronary artery disease [Count of Participants; unit: Participants]
  Yes | 21 | 383 | 404
  No | 98 | 2547 | 2645

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved >5% Weight Loss at 12 Months
Description: Participants who had both a baseline and 12 month weight measurement were included. Weight change at 12 months was measured as a percent difference from their starting weight.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Intervention Group: Subjects who were offered the toolbox of weight loss interventions and paid at least one co-pay to start using a tool. Included in analysis if they had both baseline and 12 month weights available.
- Registry-Based Control Group: Eligible subjects from an obesity registry (i.e. BMI >/= 30 and at least one weight-related comorbidity) who had at least one measured weight during usual care during the 12-month study period. Included in analysis if they had both baseline and 12 month weights available.
Arm/Group | Intervention Group | Registry-Based Control Group
Number analyzed (Participants) | 113 | 2640
percentage of participants | 34.5 | 15.7
Statistical Analysis 1: Comparison: Intervention Group vs Registry-Based Control Group; Test type: Other; p < 0.001, Chi-squared

2. Primary Outcome: Health Care Utilization - Non-study Clinic Visits
Description: Evaluation of differences in health care resource utilization between Tool and Control groups during the study period. Health care resource utilization defined as the number of non-study clinic visits.
Time Frame: 1 year study period
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of visits
Arm/Group | Intervention Group | Registry-Based Control Group
Number analyzed (Participants) | 119 | 2930
Number of visits | 4.44 [3.89 to 5.06] | 4.32 [4.20 to 4.43]

3. Secondary Outcome: Documentation of Obesity
Description: To assess:
  1. Presence of ICD-9 code for obesity in the DHHA registry Control Group
  2. Evidence of a specific intervention for weight management resembling what was offered in the toolbox intervention: weight loss medication prescribed, gym membership, weight loss program or referral to wt loss specialist, and meal replacements
Time Frame: 1 year study period
Population: Random sample of 120 patient medical records from the DHHA registry Control Group with recorded BMI > or = to 30 plus one comorbidity
Measure: Count of Participants; unit: Participants
Groups:
- Random Sample of DHHA Registry Control Group: We selected a random sample of 120 patients from the DHHA registry Control Group for a chart review. The dates used matched the study intervention period. Six reviewers, 3 MDs and 3 study personnel, reviewed medical records for the following:
  1. Presence of ICD-9 code for obesity
  2. Evidence that the the PCP discussed weight loss with the patient
  3. Evidence of a specific intervention for weight management. Each record was evaluated by two reviewers, 1 MD and 1 study personnel .
Arm/Group | Random Sample of DHHA Registry Control Group
Number analyzed (Participants) | 120
Participants
  ICD-Code for Obesity in Chart: Present | 52
  ICD-Code for Obesity in Chart: Absent | 68
  Specific Intervention provided: Present | 14
  Specific Intervention provided: Absent | 106

4. Primary Outcome: Health Care Utilization - Laboratory Measurements
Description: Evaluation of differences in health care resource utilization between Tool and Control groups during the study period. Health care resource utilization defined as the number of number of lab measurements taken during the period (including A1C, creatinine, and lipids).
Time Frame: 1 year study period
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of measurements
Arm/Group | Intervention Group | Registry-Based Control Group
Number analyzed (Participants) | 119 | 2930
Number of measurements
  A1C measurements | 1.19 [1.01 to 1.41] | 1.19 [1.15 to 1.23]
  Creatinine measurements | 2.17 [1.71 to 2.74] | 2.20 [2.10 to 2.31]
  Lipid measurements | 0.45 [0.34 to 0.58] | 0.41 [0.39 to 0.43]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the first patient in the intervention arm received a tool at their study visit #1 (1/14/2015) through when the final study patient was seen for receiving a tool at their study visit #12 (8/12/2016). Thus, adverse events were collected over a period of 19 months. Adverse events were not collected on those in the control arm; those subjects participated passively by a waiver of consent and never had any interaction with the study team.
Description: The definitions used by clinicaltrials.gov for adverse event and serious adverse event apply. Adverse events were only collected and reported on the intervention arm only and not on the control arm, as those in the control participated passively by a waiver of consent and never had any interaction with the study team or knowledge of the study's existence. This waiver was approved by the IRB.
Groups:
- Intervention: 428 randomly-selected patients from four Denver Health clinics were selected to be offered a "toolbox" of weight loss options, including: self-monitoring tools; education materials; recreation center passes; commercial weight loss program vouchers (Weight Watchers); intensive group counseling (Colorado Weigh); meal replacements (shakes & entrees); and obesity pharmacotherapy (Qsymia & phentermine) for a $5-$10 co-pay for the therapies. Of these 428 patients, 140 came in and consented at the computer program visit at which these options were offered. 119 of these patients came in for a visit one where they received their tool for the first time. Adverse events from the group of 140 patients who consented to receive the intervention are reported.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 1/140
Serious Adverse Events (participants affected / at risk) | 1/140
Other Adverse Events (participants affected / at risk) | 9/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=140)
Death occurring after being lost to follow up for a year on meal replacement tool (General disorders) | 1 (1) — After being lost-to-follow-up for 1 year after 1 visit where meal replacements were dispensed, study staff learned tyring to follow up for final feedback visit that patient had passed away. The PI, IRB, and Sponsor determined his death was unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=140)
Fainting on Qsymia (General disorders) | 1 (1) — Fainting on Qsymia (study medication tool used in routine clinical care); classified as other adverse event, not SAE
Depression on Qsymia (Psychiatric disorders) | 1 (1) — Depression on Qsymia (medication tool in the study used in routine clinical care); classified as other adverse event, not SAE
Anxiety/Chest Pain on Qsymia (Psychiatric disorders) | 1 (1) — Anxiety/Chest Pain on Qsymia; (medication tool used in routine clinical care); classified as other adverse event, not SAE
GERD causing chest pain on Qsymia (Gastrointestinal disorders) | 1 (1) — GERD causing chest pain on Qsymia;( medication tool used in routine clinical care); classified as other adverse event, not SAE
Unknown chest pain on Qsymia (General disorders) | 1 (1) — Unknown chest pain on Qsymia; (medication tool used in routine clinical care); classified as other adverse event, not SAE
Eye pain on Qsymia (Eye disorders) | 1 (1) — Eye pain on Qsymia; (medication tool used in routine clinical care); classified as other adverse event, not SAE
CVA (stroke) on Weight Watchers (Vascular disorders) | 1 (1) — CVA (stroke) on Weight Watchers; one of the study tools available that would be determined as unrelated to stroke; classified as other adverse event, not SAE
Alcohol withdrawal symptoms (General disorders) | 2 (2) — Alcohol withdrawal symptoms; unrelated to study tool or procedures; classified as other adverse event, not SAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less